CLINICAL TRIAL: NCT07087340
Title: Early Feasibility Evaluation of the UniBE Hybrid Closed-loop Insulin Delivery System in Type 1 Diabetes: UBLoop - Genesis
Brief Title: Early Feasibility Evaluation of the UniBE Hybrid Closed-loop Insulin Delivery System in Type 1 Diabetes: UBLoop-Genesis
Acronym: UBLoop-Gen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: DCB Research AG (Other); DexCom, Inc. (Industry); mylife Diabetes Care AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025-D0056
Record Dates: First submitted 2025-07-24; First posted 2025-07-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Type-1-Diabetes
Keywords: Automated insulin delivery; Artificial pancreas

STUDY DESIGN:
Intervention Model Description: Single-center, single-arm, supervised study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UBLoop Intervention Group (Experimental): For a period of approximately 10 hours, study participants will wear an insulin pump and a continuous glucose monitor (CGM), with the UBLoop system controlling insulin delivery based on the CGM readings. The UBLoop system will be operating via an app installed on a smartphone.
  Interventions: Device: UBLoop System

INTERVENTIONS:
Device: UBLoop System — Participants (people living with Type-1-Diabetes) will attend a study visit where the UBLoop system will manage insulin delivery via an insulin pump, using blood glucose values from a continuous glucose meter (CGM). Specialized staff and a remote monitoring system, which is integrated into the UBLoop system, will oversee the participants. The investigational product comprises (1) the BernSHELL App, communicating with the CGM and the insulin pump, (2) the UBLoop algorithm receiving CGM data, processing the control algorithm, calculating insulin dosing, checking the safety of the calculated insulin injections, and transmitting instructions to the insulin pump via BernSHELL, (3) the UBLoop Cloud providing secure storage, analytics support, and data backup, (4) DigiCare, monitoring the safety of the study participants and the system's execution flow in real time.
  During the intervention, participants will use the Ypsomed myLife YpsoPump (insulin pump) and the Dexcom G6 or G7 CGM.

SUMMARY:
The study is investigating the early feasibility of a novel algorithm for a hybrid closed-loop (HCL) insulin delivery system in adult patients with Type 1 diabetes.

Participants will attend a study visit where the UBLoop system on a smartphone will manage insulin delivery via an insulin pump, using blood glucose values from a continuous glucose meter. Specialized staff and a remote monitoring system, which is integrated into the UBLoop system, will oversee the participants.

ELIGIBILITY:
Inclusion Criteria:

* T1D diagnosis for at least one year.
* Aged between 18 and 65 years old (inclusive).
* Currently using insulin for at least six months.
* Currently using closed-loop insulin therapy for at least three months.
* Willingness to suspend any personal CGM for the duration of the pilot study once the study CGM is in place.
* Willingness not to start any new non-insulin glucose-lowering agent during the study (including metformin/biguanides, incretin agonists [GIP/GLP-1RAs or GLP-1RAs], pramlintide, DPP-4 inhibitors, sulfonylureas, Sodium-glucose cotransporter-2 inhibitors [SGLT2 inhibitors], and nutraceuticals).
* Understanding and willingness to follow the protocol and signed informed consent.

Exclusion Criteria:

* An HbA1C ≥10% .
* History of diabetic ketoacidosis (DKA) in the past 12 months.
* History of severe hypoglycaemic event (Level 3): defined as seizure or loss of consciousness in the past 12 months.
* Current uncontrolled chronic diabetic microvascular complications (neuropathy, retinopathy, renal diabetes disease, and diabetic gastroparesis).
* Body Mass Index (BMI) ≤18.5 or ≥ 35 kg m2
* Estimated glomerular filtration rate (eGFR) lab value below 30 mL/min/1.73 m2
* Pregnancy or intent to become pregnant during the study.
* Currently breastfeeding or planning to breastfeed.
* Currently uncontrolled seizure disorder.
* Planned surgery during the study duration.
* Have uncontrolled hypertension (systolic BP above or equal to 160 mmHg and/or diastolic BP above or equal to 100 mmHg). If a participant is on anti-hypertensive therapies, doses must be stable for 30 days before screening. For participants with uncontrolled hypertension at the screening visit, antihypertensive medication may be started or adjusted.*
* Personal history of one of the following cardiovascular conditions: acute myocardial infarction, cerebrovascular accident (stroke), unstable angina, or hospitalization due to congestive heart failure (CHF) in the last three months before the screening.
* Conditions that may increase the risk of induced hypoglycemia such as known coronary artery disease, CHF (Have NYHA Functional Classification III or IV CHF), history of any cardiac disorder or arrhythmia, history of cerebrovascular event, hypoglycemia-induced migraine within the past six months, seizure disorder, syncope, adrenal insufficiency, or neurological disease).
* Cystic fibrosis.
* Uncontrolled thyroid disease as judged by the investigator.
* Have an uncontrolled psychiatric condition such as (major depressive disorder, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder, alcohol or drug abuse).
* Treatment with a non-insulin glucose-lowering agent, except metformin, in stable doses in the last three months.
* Participants receiving or have received systemic glucocorticoid therapy within three months before screening (Prednisolone 10mg daily or equivalent >2 weeks) or chronic systemic glucocorticoid therapy (excluding topical, intraocular, intranasal, single intraarticular injection, or inhaled preparations).
* Have current treatment with (or history of, within 3 months before screening) medications that may affect glucose metabolism, as judged by the investigator.
* Current enrolment in another clinical trial, unless approved by the investigator of both studies, and if the clinical trial is a non-interventional registry trial.
* Have evidence of a significant active, uncontrolled medical condition or a history of any medical problem capable of constituting a risk when using the study devices or interfering with the interpretation of data, as judged by the study physician at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of time with the system functioning in closed-loop mode | 10 hours
Failure rate of the HCL algorithm | 10 hours
Failure rate of the communication with CGM device | 10 hours
Failure rate of the communication with Insulin pump | 10 hours
Failure rate of the user interface (BernSHELL) | 10 hours
Failure rate of the web monitoring tool (DigiCARE) | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, Prof.Dr.med., Principal Investigator — Universitätsklinik für Diabetologie, Endokrinologie, Ernährungsmedizin & Metabolismus (UDEM)
Locations (1):
- Inselspital, Universitätsspital; Universitätsklinik für Diabetologie, Endokrinologie, Ernährungsmedizin & Metabolismus (UDEM), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No